CLINICAL TRIAL: NCT01244490
Title: A Phase 3, Randomised, Double-blind, Multicentre, Parallel-group, Placebo- and Active-reference, Dose-optimisation Efficacy and Safety Study of Extended-release Guanfacine Hydrochloride in Children and Adolescents Aged 6-17 Years With Attention-Deficit/Hyperactivity Disorder
Brief Title: Efficacy and Safety of Extended-release Guanfacine Hydrochloride in Children and Adolescents Aged 6-17 Years With Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPD503-316; 2010-018579-12 (EudraCT Number)
Record Dates: First submitted 2010-11-16; First posted 2010-11-19 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Guanfacine; Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Extended-release Guanfacine Hydrochloride (Experimental)
  Interventions: Drug: Extended-release Guanfacine Hydrochloride
- Atomoxetine Hydrochloride (Other): Active Reference
  Interventions: Drug: Atomoxetine Hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Extended-release Guanfacine Hydrochloride — Tablet, once daily, optimised dose (1mg to 7mg based on age and weight), 6-week maintenance duration on optimised dose.
  Other Names: Intuniv
  Arms: Extended-release Guanfacine Hydrochloride
Drug: Atomoxetine Hydrochloride — Capsule, once daily, optimised dose (10mg to 100mg based on weight), 8-9-weeks maintenance duration on optimised dose
  Other Names: Strattera
  Arms: Atomoxetine Hydrochloride
Drug: Placebo Comparator — Placebo
  Arms: Placebo

SUMMARY:
For children and adolescents, how does SPD503 compare to placebo for the treatment of Attention-Deficit/Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 6 17 years at the time of consent/assent at Screening (Visit 1).
2. Subject's parent or legally authorised representative (LAR) must provide signature of informed consent, and there must be documentation of assent (if applicable) by the subject indicating that the subject is aware of the investigational nature of the study and the required procedures and restrictions in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guidance E6, and applicable regulations before completing any study related procedures at Screening (Visit 1).
3. Subject meets Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria for a primary diagnosis of ADHD, combined sub-type, hyperactive/impulsive sub-type, or inattentive sub-type based on a detailed psychiatric evaluation using the Kiddie Schedule for Affective Disorders and Schizophrenia - Present and Lifetime version (K-SADS-PL).
4. Subject has a minimum ADHD-RS-IV total score of 32 at Baseline (Visit 2).
5. Subject has a minimum CGI-S score of 4 at Baseline (Visit 2).
6. Subject is functioning at an age-appropriate level intellectually, as judged by the Investigator.
7. Subject and parent/LAR understand, are willing, able, and likely to fully comply with the study procedures and restrictions defined in this protocol.
8. Subject is able to swallow intact tablets and capsules.
9. Subject who is a female of child-bearing potential (FOCP), defined as greater than or equal to 9 years of age or <9 years of age and is menarchal, must have a negative serum beta Human Chorionic Gonadotropin (hCG) pregnancy test at Screening (Visit 1) and a negative urine pregnancy test at Baseline (Visit 2) and agree to comply with any applicable contraceptive requirements of the protocol.
10. Subject has supine and standing blood pressure (BP) measurement within the 95th percentile for age, sex, and height

Exclusion Criteria:

1. Subject has a current, controlled (requiring a prohibited medication or behavioural modification program) or uncontrolled, co-morbid psychiatric diagnosis [except oppositional defiant disorder (ODD)], including any severe co-morbid Axis II disorders or severe Axis I disorders such as post traumatic stress disorder (PTSD), bipolar illness, psychosis, pervasive developmental disorder, obsessive-compulsive disorder (OCD), substance abuse disorder, or other symptomatic manifestations or lifetime history of bipolar illness, psychosis or conduct disorder that, in the opinion of the Investigator, contraindicate treatment with SPD503 or STRATTERA or confound efficacy or safety assessments.
2. Subject is well-controlled on their current medication, with acceptable tolerability, and the parent/caregiver does not object to the current medication.
3. Subject has any condition or illness including a clinically significant abnormal Screening (Visit 1) laboratory values which, in the opinion of the Investigator, represents an inappropriate risk to the subject and/or could confound the interpretation of the study. Mild stable asthma treated without the use of beta-2 agonist is not exclusionary.
4. Subject has a known history or presence of structural cardiac abnormalities, cardiovascular or cerebrovascular disease, serious heart rhythm abnormalities, syncope, tachycardia, cardiac conduction problems (eg, clinically significant heart block or QT interval prolongation), exercise-related cardiac events including syncope and pre syncope, or clinically significant bradycardia.
5. Subject has a known family history of sudden cardiac death, ventricular arrhythmia, or QT prolongation.
6. Subjects with orthostatic hypotension or a known history of hypertension.
7. Subject has glaucoma.
8. Subject has clinically significant ECG findings as judged by the Investigator with consideration of the central ECG laboratory's interpretation.
9. Subject has a history of a seizure disorder (other than a single childhood febrile seizure occurring before the age of 3 years) or the presence of a serious tic disorder including Tourette's Syndrome.
10. Current use of any prohibited medication or other medications, including monoamine oxidase inhibitors, herbal supplements, that affect BP or heart rate potent CYP2D6 inhibitors, medications known to prolong the QT/QTc interval, medications that lower seizure threshold, pressor agents, beta-2 agonists, medications that affect noradrenaline, medications that have central nervous system (CNS) effects or affect cognitive performance, such as sedating antihistamines and decongestant sympathomimetics (inhaled bronchodilators are permitted) or a history of chronic use of sedating medications [ie, antihistamines]) in violation of the protocol specified washout criteria at Baseline (Visit 2).
11. Subject has a history of alcohol or other substance abuse or dependence, as defined by DSM-IV (with the exception of nicotine) within the last 6 months.
12. Subject has taken another investigational product within 30 days prior to Baseline (Visit 2).
13. Subject is significantly overweight based on Center for Disease Control and Prevention Body Mass Index (BMI)-for-age gender specific charts at the Screening (Visit 1). Significantly overweight is defined as a BMI >95th percentile.
14. Children aged 6 12 years with a body weight of less than 25kg or adolescents aged 13 17 years with a body weight of less than 34kg or greater than 91kg at Screening (Visit 1).
15. Subject has a known or suspected allergy, hypersensitivity, or clinically significant intolerance to guanfacine hydrochloride or atomoxetine hydrochloride, or any components found in SPD503 or STRATTERA.
16. Clinically important abnormality on drug and alcohol screen (excluding the subject's current ADHD stimulant if applicable) at Screening (Visit 1)
17. Subject is female and is pregnant or currently lactating.
18. Subject failed screening or was previously enrolled in this study.
19. Subject is currently considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating active suicide ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the Investigator.
20. History of failure to respond to an adequate trial of an α2-agonist or atomoxetine hydrochloride for the treatment of ADHD (consisting of an appropriate dose and adequate duration of therapy in the opinion of the investigator).
21. Subjects with renal or hepatic insufficiency.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 338 (Actual)
Dates: Start 2011-01-17 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (66):
- United States (11):
  - Psychiatric Centers at San Diego, Feighner Research, San Diego, California
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Psychiatric Associates, Overland Park, Kansas
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - University of Nebraska Medical Center, Dept. of Psychiatry, Omaha, Nebraska
  - Innovis Health, Fargo, North Dakota
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - Claghorn-Lesem Research Clinic, Houston, Texas
  - R/D Clincial Research, Inc., Lake Jackson, Texas
  - NeuroScience Inc., Herndon, Virginia
- Austria (2):
  - Medizinische Universitat Graz-Universitaklinik fur Kinder-und Jugendheilkunde, Graz
  - Institut für Psychosomatik, Vienna
- Canada (2):
  - Dr Grazyna B. Jackiewicz, MD, Niagara Falls, Ontario
  - JPM Van Stralen Medicine Professional Corp., Ottawa, Ontario
- France (3):
  - Centre HospitalierUniversitaire d'Amiens, Hoptial Nord, Amiens, Picardie
  - Centre Hospitalier Charles Perens - Service de Psychiatrie de l'Enfant et de l'Adolescent, Bordeaux
  - Centre Hospitalier des Pyrenees, Chartres
- Germany (11):
  - Praxis Dr. Wolff, Hagen, North Rhine-Westphalia
  - Praxis Dr. Andreas Mahler, Achim
  - Emovis GmbH, Berlin
  - Universitaetsklinikum Carl Gustav Carus an der Technischen Universitaet Dresden, Dresden
  - Praxisgemeinschaft Drs. Willem Geraets/Gabriele Lucassen, Düsseldorf
  - Praxis Dr. Walter Robert Otto, Fulda
  - Praxis Dr. Friedrich Kaiser un Ingrid Marinesse, Hamburg
  - Institut fur Ganzheitiche Medzin und Wissenschaft GmbH, Hüttenberg
  - Klinikum der Johannes-Guttenberg-Universitat Mainz, Mainz
  - Zentralinstitut fur Seelische Geseundheit Mannheim Klinik for Psuchiatrie und Psychotherapie des Kindes, Mannheim
  - Somni Bene GmbH - Institut für Medizinische Forschung und Schlafmedizin, Schwerin
- Department of Child and Adolescent Psychiatry, Dublin, Ireland
- Italy (3):
  - IRCCS Stella Maris - U.O. Psichiatria e Psicofarmacologia Eta' Evolutiva, Pisa
  - Università Cattolica del Sacro Cuore, Rome
  - Ospedale Policlinico G.B.Rossi - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Poland (6):
  - Indywidualna Specjalistyczna Praktyka Lekarska Borys Gniot, Torun, Kuyavian-Pomeranian Voivodeship
  - Centrum Neuropsychiatrii Neuromed, Wroclaw, Lower Silesian Voivodeship
  - Samodzielny Publiczny Dzieciecy Szpital Kliniczny, Warsaw, Masovian Voivodeship
  - Centrum Badan Klinicznych PI-House Sp. z o.o., Gdansk, Pomeranian Voivodeship
  - NZOZ Gdan Skie Centrum Zdrowia, Gdansk
  - Gabinet Psychiatrii Doroslych, Dzieci i Mlodziezy, Miroslaw Dabkowski, Torun
- Romania (4):
  - Spitalul Clinic de Urgenta Pentru Copii Cluj, Cluj-Napoca, Cluj
  - Spitalul Clinic de Urgenta pentru Copii "Louis Turcanu", Timișoara, Timiș County
  - Spitalul Clinic de Psihiatrie "Prof. Dr. Alexandru Obregia", Bucharest
  - Spitalul Clinic de Psihiatrie Socola, Iași
- Spain (7):
  - Mutua de Terrassa, Terrassa, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Policlínica Guipuzkoa, Donostia / San Sebastian
  - Hospital Marítimo, (USMI-J), Málaga
  - Hospital de Dia Infantil y Juvenil Dr Diego Guigou y Costa, Santa Cruz de Tenerife
  - Hospital Universitario Marques de Valdecilla, Santander
  - Instituto Valenciano de Neurología Pediatrica, Valencia
- Sweden (3):
  - Drottning Silvias Barnsjukhus, Gothenburg
  - Barn och Ungdomsmedicin klinik Mölnlycke, Mölnlycke
  - BUP mottagningen Varberg, Varberg
- Ukraine (8):
  - Institute of Neurology, Psychiatry and Narcology of the AMS of Ukraine, Kharkiv, Kharkivs’ka Oblast’
  - Regional Clinical Psychiatric Hospital, Donetsk
  - Municipal Institution "Institute of healthcare for children and adolescences NAMNU, Kharkiv
  - Kherson Regional Psychiatric Hospital, Kherson
  - Lviv Regional Clinical Psychiatric Hospital, Lviv
  - Odesa Regional Psychoneurological Dispensary, Outpatient Dept, Odesa
  - O.F. Maltsev Poltava Regional Psychiatric Hospital, Poltava
  - Vinnytsia National Medical University - Vinnytsia Regional Psycho-Neurological Hospital, Vinnytsia
- United Kingdom (5):
  - Victoria Hospital, Kirkcaldy, Fife
  - James Paget University Hospital NHS Trust, Great Yarmouth, Norfolk
  - Ashurt Child and Family Centre, Ashurst, Southampton
  - Horsham Child and Adolescent Mental Health Services, Horsham
  - 5 Boroughs Partnership NHS Trust, Wigan

REFERENCES:
- [Result] Hervas A, Huss M, Johnson M, McNicholas F, van Stralen J, Sreckovic S, Lyne A, Bloomfield R, Sikirica V, Robertson B. Efficacy and safety of extended-release guanfacine hydrochloride in children and adolescents with attention-deficit/hyperactivity disorder: a randomized, controlled, phase III trial. Eur Neuropsychopharmacol. 2014 Dec;24(12):1861-72. doi: 10.1016/j.euroneuro.2014.09.014. Epub 2014 Oct 23. PMID 25453486

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Once daily
- Guanfacine Hydrochloride: Tablet, once daily, optimised dose (1mg to 7mg based on age and weight)
- Atomoxetine Hydrochloride: Capsule, once daily, optimised dose (10mg to 100mg based on weight)
Period: Overall Study
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Started | 111 | 115 | 112
Completed | 92 | 91 | 89
Not Completed | 19 | 24 | 23
Not completed — Lack of Efficacy | 14 | 5 | 5
Not completed — Withdrawal by Subject | 4 | 4 | 9
Not completed — Adverse Event | 1 | 9 | 5
Not completed — Lost to Follow-up | 0 | 6 | 3
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population defined as all randomized subjects who took at least 1 dose of investigational product. One subject did not receive investigational product, therefore n = 337.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride | Total
Number analyzed (Participants) | 111 | 114 | 112 | 337
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.0 (2.76) | 10.9 (2.77) | 10.5 (2.81) | 10.8 (2.78)
Age, Customized [Count of Participants; unit: Participants]
  6-12 years | 79 | 81 | 82 | 242
  13-17 years | 32 | 33 | 30 | 95
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 38 | 25 | 88
  Male | 86 | 76 | 87 | 249
Region of Enrollment [Count of Participants; unit: Participants]
  AUSTRIA | 2 | 4 | 5 | 11
  CANADA | 6 | 7 | 6 | 19
  FRANCE | 2 | 2 | 2 | 6
  GERMANY | 23 | 23 | 22 | 68
  IRELAND | 0 | 1 | 1 | 2
  ITALY | 5 | 4 | 4 | 13
  POLAND | 11 | 14 | 12 | 37
  ROMANIA | 5 | 3 | 6 | 14
  SPAIN | 16 | 18 | 17 | 51
  SWEDEN | 1 | 1 | 2 | 4
  UKRAINE | 21 | 18 | 15 | 54
  UNITED KINGDOM | 1 | 0 | 1 | 2
  UNITED STATES | 18 | 19 | 19 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale-fourth Edition (ADHD-RS-IV) Total Score at Week 10/13 - Last Observation Carried Forward (LOCF)
Description: The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54. Outcome measure is at 10 weeks for ages 6-12 years and at 13 weeks for ages 13-17 years.
Time Frame: Baseline and Up to 10 weeks for children aged 6-12 years and up to 13 weeks for adolescents aged 13-17 years
Population: Full Analysis Set (FAS) defined as all randomized subjects who took at least 1 dose of investigational product. If more than 20% of the items used for summing a score were missing, the score was set to missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 111 | 112 | 112
units on a scale | -15.0 (1.1612) | -23.9 (1.1531) | -18.8 (1.1549)
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in Least Squares Mean = -8.9, 95% CI 2-sided [-11.9 to -5.8]
Statistical Analysis 2: Comparison: Placebo vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.017, ANCOVA; Difference in Least Squares Mean = -3.8, 95% CI 2-sided [-6.8 to -0.7]

2. Secondary Outcome: Percentage of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I) Scores
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale. Outcome measure is at 10 weeks for ages 6-12 years and at 13 weeks for ages 13-17 years.
Time Frame: Up to 10 weeks for children aged 6-12 years and up to 13 weeks for adolescents aged 13-17 years
Population: Full Analysis Set. Not all subjects in the FAS population had data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 111 | 112 | 112
percentage of participants | 44.1 | 67.9 | 56.3
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Difference in Percentage Improvement = 23.7, 95% CI 2-sided [11.1 to 36.4]
Statistical Analysis 2: Comparison: Placebo vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.024, Cochran-Mantel-Haenszel; Difference in Percentage Improvement = 12.1, 95% CI 2-sided [-0.9 to 25.1]

3. Secondary Outcome: Change From Baseline in the Weiss Functional Impairment Rating Scale - Parent Report (WFIRS-P) Learning and School Domain Scores at Week 10/13 - LOCF
Description: The WFIRS-P Learning in School Domain is the mean of 10 items, ranging from 0 (never/not at all) to 3 (very often/very much). Higher scores indicate greater functional impairment. Outcome measure is at 10 weeks for ages 6-12 years and at 13 weeks for ages 13-17 years.
Time Frame: Baseline and Up to 10 weeks for children aged 6-12 years and up to 13 weeks for adolescents aged 13-17 years
Population: Full Analysis Set. If more than 30% of items used to derive the score were missing, the corresponding score was considered as missing.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 100 | 103 | 100
units on a scale | -0.419 (0.0537) | -0.636 (0.0527) | -0.581 (0.0534)
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p = 0.003, ANCOVA; Difference in Least Squares Mean = -0.217, 95% CI 2-sided [-0.358 to -0.076]
Statistical Analysis 2: Comparison: Placebo vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.026, ANCOVA; Difference in Least Squares Mean = -0.162, 95% CI 2-sided [-0.305 to -0.019]

4. Secondary Outcome: Change From Baseline in the WFIRS-P Family Domain Score at Week 10/13 - LOCF
Description: The WFIRS-P Family Domain is the mean of 10 items, ranging from 0 (never/not at all) to 3 (very often/very much). Higher scores indicate greater functional impairment. Outcome measure is at 10 weeks for ages 6-12 years and at 13 weeks for ages 13-17 years.
Time Frame: Baseline and Up to 10 weeks for children aged 6-12 years and up to 13 weeks for adolescents aged 13-17 years
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 106 | 109 | 105
units on a scale | -0.409 (0.0568) | -0.617 (0.0558) | -0.499 (0.0566)
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p = 0.006, ANCOVA; Difference in Least Squares Mean = -0.209, 95% CI 2-sided [-0.358 to -0.059]
Statistical Analysis 2: Comparison: Placebo vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.242, ANCOVA; Difference in Least Squares Mean = -0.090, 95% CI 2-sided [-0.241 to 0.061]

5. Secondary Outcome: Clinical Global Impression-Severity of Illness (CGI-S) - LOCF
Description: CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill). Outcome measure is at 10 weeks for ages 6-12 years and at 13 weeks for ages 13-17 years.
Time Frame: Up to 10 weeks for children aged 6-12 years and up to 13 weeks for adolescents aged 13-17 years
Population: Full Analysis Set. Not all subjects in the FAS population had data for this outcome.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 111 | 112 | 112
percentage of participants
  1 (Normal, not at all ill) | 9.9 | 14.3 | 6.3
  2 (Borderline mentally ill) | 15.3 | 23.2 | 19.6
  3 (Mildly ill) | 20.7 | 31.3 | 32.1
  4 (Moderately ill) | 20.7 | 22.3 | 19.6
  5 (Markedly ill) | 25.2 | 5.4 | 13.4
  6 (Severely ill) | 6.3 | 3.6 | 7.1
  7 (Amongst the most extremely ill) | 1.8 | 0 | 1.8
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Nominal p-value uncorrected for multiplicity
Statistical Analysis 2: Comparison: Placebo vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.196, Cochran-Mantel-Haenszel — Nominal p-value uncorrected for multiplicity

6. Secondary Outcome: Health Utilities Index-2/3 (HUI 2/3) Scores - LOCF
Description: HUI is used to describe health status and to obtain utility scores by collecting data using one or more questionnaires in formats selected to match the specific study design criteria. Scoring ranges from 0.00 (dead) to 1.00 (perfect health). Higher scores represent better health status. Outcome measure is at 10 weeks for ages 6-12 years and at 13 weeks for ages 13-17 years.
Time Frame: Up to 10 weeks for children aged 6-12 years and up to 13 weeks for adolescents aged 13-17 years
Population: Full Analysis Set. Not all subjects in the FAS population had data for this outcome.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 106 | 110 | 106
units on a scale | 0.927 (0.0950) | 0.922 (0.0908) | 0.913 (0.1052)

7. Secondary Outcome: Change From Baseline in the WFIRS-P Global Score at Week 10/13 - LOCF
Description: The WFIRS-P Global Score is the mean of 50 items, ranging from 0 (never/not at all) to 3 (very often/very much). Higher scores indicate greater functional impairment. Outcome measure is at 10 weeks for ages 6-12 years and at 13 weeks for ages 13-17 years.
Time Frame: Baseline and Up to 10 weeks for children aged 6-12 years and up to 13 weeks for adolescents aged 13-17 years
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 104 | 110 | 104
units on a scale | -0.321 (0.0387) | -0.487 (0.0374) | -0.425 (0.0384)
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p = 0.001, ANCOVA — Nominal p-value uncorrected for multiplicity; Mean Difference (Final Values) = -0.165, 95% CI 2-sided [-0.266 to -0.064]
Statistical Analysis 2: Comparison: Placebo vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.048, ANCOVA — Nominal p-value uncorrected for multiplicity; Mean Difference (Final Values) = -0.104, 95% CI 2-sided [-0.207 to -0.001]

8. Secondary Outcome: Change From Baseline in the WFIRS-P Academic Performance Domain Score at Week 10/13 - LOCF
Description: The WFIRS-P Academic Performance Domain is the mean of 4 items, ranging from 0 (never/not at all) to 3 (very often/very much). Higher scores indicate greater functional impairment. Outcome measure is at 10 weeks for ages 6-12 years and at 13 weeks for ages 13-17 years.
Time Frame: Up to 10 weeks for children aged 6-12 years and up to 13 weeks for adolescents aged 13-17 years
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 96 | 103 | 101
units on a scale | -0.555 (0.0784) | -0.766 (0.0757) | -0.681 (0.0759)
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p = 0.043, ANCOVA — Nominal p-value uncorrected for multiplicity; Difference in Least Squares Mean = -0.211, 95% CI 2-sided [-0.416 to -0.007]
Statistical Analysis 2: Comparison: Placebo vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.231, ANCOVA — Nominal p-value uncorrected for multiplicity; Difference in Least Squares Mean = -0.125, 95% CI 2-sided [-0.331 to 0.080]

9. Secondary Outcome: Change From Baseline in the WFIRS-P Behavior in School Domain Score at Week 10/13 - LOCF
Description: The WFIRS-P Behavior in School Domain is the mean of 6 items, ranging from 0 (never/not at all) to 3 (very often/very much). Higher scores indicate greater functional impairment. Outcome measure is at 10 weeks for ages 6-12 years and at 13 weeks for ages 13-17 years.
Time Frame: Up to 10 weeks for children aged 6-12 years and up to 13 weeks for adolescents aged 13-17 years
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 100 | 103 | 100
units on a scale | -0.363 (0.0512) | -0.592 (0.0502) | -0.544 (0.0509)
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p < 0.001, ANCOVA — Nominal p-value uncorrected for multiplicity; Diiference in Least Squares Mean = -0.229, 95% CI 2-sided [-0.364 to -0.094]
Statistical Analysis 2: Comparison: Placebo vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.009, ANCOVA — Nominal p-value uncorrected for multiplicity; Difference in Least Squares Mean = -0.181, 95% CI 2-sided [-0.317 to -0.045]

10. Secondary Outcome: Change From Baseline in the WFIRS-P Life Skills Domain Score at Week 10/13 - LOCF
Description: The WFIRS-P Life Skills Domain is the mean of 10 items, ranging from 0 (never/not at all) to 3 (very often/very much). Higher scores indicate greater functional impairment. Outcome measure is at 10 weeks for ages 6-12 years and at 13 weeks for ages 13-17 years.
Time Frame: Up to 10 weeks for children aged 6-12 years and up to 13 weeks for adolescents aged 13-17 years
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 105 | 110 | 104
units on a scale | -0.383 (0.0422) | -0.477 (0.0411) | -0.450 (0.0422)
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p = 0.096, ANCOVA — Nominal p-value uncorrected for multiplicity; Difference in Least Squares Mean = -0.094, 95% CI 2-sided [-0.204 to 0.017]
Statistical Analysis 2: Comparison: Placebo vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.242, ANCOVA — Nominal p-value uncorrected for multiplicity; Difference in Least Squares Mean = -0.067, 95% CI 2-sided [-0.180 to 0.046]

11. Secondary Outcome: Change From Baseline in the WFIRS-P Child Self-Concept Domain Score at Week 10/13 - LOCF
Description: The WFIRS-P Child Self-Concept Domain is the mean of 3 items, ranging from 0 (never/not at all) to 3 (very often/very much). Higher scores indicate greater functional impairment. Outcome measure is at 10 weeks for ages 6-12 years and at 13 weeks for ages 13-17 years.
Time Frame: Up to 10 weeks for children aged 6-12 years and up to 13 weeks for adolescents aged 13-17 years
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 101 | 108 | 103
units on a scale | -0.312 (0.0544) | -0.361 (0.0528) | -0.390 (0.0536)
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p = 0.500, ANCOVA — Nominal p-value uncorrected for multiplicity; Difference in Least Squares Mean = -0.049, 95% CI 2-sided [-0.191 to 0.094]
Statistical Analysis 2: Comparison: Placebo vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.288, ANCOVA — Nominal p-value uncorrected for multiplicity; Difference in Least Squares Mean = -0.078, 95% CI 2-sided [-0.222 to 0.066]

12. Secondary Outcome: Change From Baseline in the WFIRS-P Social Domain Score at Week 10/13 - LOCF
Description: The WFIRS-P Social Domain is the mean of 7 items, ranging from 0 (never/not at all) to 3 (very often/very much). Higher scores indicate greater functional impairment. Outcome measure is at 10 weeks for ages 6-12 years and at 13 weeks for ages 13-17 years.
Time Frame: Up to 10 weeks for children aged 6-12 years and up to 13 weeks for adolescents aged 13-17 years
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 104 | 110 | 104
units on a scale | -0.322 (0.0537) | -0.555 (0.0519) | -0.434 (0.0532)
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p = 0.001, ANCOVA — Nominal p-value uncorrected for multiplicity; Difference in Least Squares Mean = -0.233, 95% CI 2-sided [-0.374 to -0.092]
Statistical Analysis 2: Comparison: Placebo vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.124, ANCOVA — Nominal p-value uncorrected for multiplicity; Difference in Least Squares Mean = -0.111, 95% CI 2-sided [-0.253 to 0.031]

13. Secondary Outcome: Change From Baseline in the WFIRS-P Risk Domain Score at Week 10/13 - LOCF
Description: The WFIRS-P Risk Domain is the mean of 10 items, ranging from 0 (never/not at all) to 3 (very often/very much). Higher scores indicate greater functional impairment. Outcome measure is at 10 weeks for ages 6-12 years and at 13 weeks for ages 13-17 years.
Time Frame: Up to 10 weeks for children aged 6-12 years and up to 13 weeks for adolescents aged 13-17 years
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 99 | 105 | 97
units on a scale | -0.134 (0.0284) | -0.190 (0.0275) | -0.173 (0.0285)
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p = 0.139, ANCOVA — Nominal p-value uncorrected for multiplicity; Difference in Least Squares Mean = -0.056, 95% CI 2-sided [-0.131 to 0.018]
Statistical Analysis 2: Comparison: Placebo vs Atomoxetine Hydrochloride; Test type: Superiority or Other; p = 0.315, ANCOVA — Nominal p-value uncorrected for multiplicity; Difference in Least Squares Mean = -0.039, 95% CI 2-sided [-0.115 to 0.037]

14. Secondary Outcome: Change From Baseline in Brief Psychiatric Rating Scale for Children (BPRS-C) Total Score at Weeks 10/13 - LOCF
Description: The BPRS-C characterizes childhood behavioral and emotional symptomatology. A total of 21 items are rated on a scale from 0 (not present) to 6 (extremely severe) with a total score ranging from 0 to 126. A decrease in score indicates a reduction in psychopathology. Outcome measure is at 10 weeks for ages 6-12 years and at 13 weeks for ages 13-17 years.
Time Frame: Baseline and up to 10 weeks for children aged 6-12 years and up to 13 weeks for adolescents aged 13-17 years
Population: Safety Population defined as of randomized subjects who took at least 1 dose of investigational product.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 102 | 101 | 99
units on a scale | -5.6 (8.82) | -8.3 (8.40) | -6.5 (9.23)

15. Secondary Outcome: Structure Side-Effect Questionnaire
Description: The Structured Side-effect Questionnaire is a simple checklist of 17 side effects. The subject indicates whether a side effect has occurred since the last visit by marking 'yes' on the checklist for each of the events listed. Outcome measure is at 12 weeks for ages 6-12 years and at 15 weeks for ages 13-17 years.
Time Frame: Up to 12 weeks for children aged 6-12 years and up to 15 weeks for adolescents aged 13-17 years
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 111 | 112 | 112
participants
  Nausea | 19 | 30 | 39
  Vomiting | 11 | 7 | 25
  Diarrhea | 15 | 18 | 8
  Abdominal Pain | 26 | 45 | 42
  Decreased Appetite | 25 | 31 | 48
  Increased Appetite | 30 | 40 | 25
  Headache | 35 | 52 | 34
  Dizziness | 16 | 28 | 23
  Fatigue | 30 | 55 | 35
  Nervousnes/Anxiety | 25 | 37 | 34
  Insomnia | 19 | 32 | 24
  Somnolence | 26 | 57 | 38
  Depression | 7 | 7 | 9
  Itching | 7 | 13 | 10
  Rash | 4 | 9 | 8
  Missed Menses | 0 | 1 | 0

16. Secondary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is a semi-structured interview that captures the occurence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behaviour occurred. The assessment is done by the nature of the responses, not by a numbered scale. Outcome measure is at 12 weeks for ages 6-12 years and at 15 weeks for ages 13-17 years.
Time Frame: Up to 12 weeks for children aged 6-12 years and up to 15 weeks for adolescents aged 13-17 years
Population: SP
Measure: Number; unit: participants
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Number analyzed (Participants) | 111 | 112 | 112
participants
  Suicidal Ideation | 2 | 3 | 5
  Suicidal Behaviour | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Guanfacine Hydrochloride | Atomoxetine Hydrochloride
Serious Adverse Events (participants affected / at risk) | 1/111 | 1/114 | 0/112
Other Adverse Events (participants affected / at risk) | 62/111 | 79/114 | 67/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=111) | Guanfacine Hydrochloride (N=114) | Atomoxetine Hydrochloride (N=112)
Syncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=111) | Guanfacine Hydrochloride (N=114) | Atomoxetine Hydrochloride (N=112)
Abdominal pain (Gastrointestinal disorders) | 20 (32) | 19 (29) | 19 (31)
Abdominal pain upper (Gastrointestinal disorders) | 6 (6) | 7 (7) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 15 (18) | 10 (16) | 2 (3)
Nausea (Gastrointestinal disorders) | 11 (13) | 18 (19) | 30 (54)
Vomiting (Gastrointestinal disorders) | 8 (9) | 6 (8) | 18 (29)
Fatigue (General disorders) | 20 (22) | 29 (45) | 24 (32)
Pyrexia (General disorders) | 4 (4) | 7 (9) | 3 (4)
Nasopharyngitis (Infections and infestations) | 6 (7) | 6 (7) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 12 (23) | 15 (20) | 31 (44)
Increased appetite (Metabolism and nutrition disorders) | 9 (11) | 12 (15) | 4 (4)
Dizziness (Nervous system disorders) | 9 (9) | 14 (18) | 17 (24)
Headache (Nervous system disorders) | 27 (46) | 30 (51) | 22 (36)
Somnolence (Nervous system disorders) | 16 (18) | 50 (94) | 20 (32)
Anxiety (Psychiatric disorders) | 8 (15) | 9 (16) | 7 (18)
Insomnia (Psychiatric disorders) | 7 (7) | 13 (21) | 8 (10)
Nervousness (Psychiatric disorders) | 6 (7) | 6 (7) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.